CLINICAL TRIAL: NCT02825108
Title: Evaluation the Effect of Intrauterine Injection of Human Chorionic Gonadotropin Injection (hCG) Before Frozen Embryo Transfer on Implantation and Clinical Pregnancy Rates Per Cycle , Phase 3 Randomized Double Blinded Clinical Trial
Brief Title: Intrauterine Injection of Human Chorionic Gonadotropin Injection (hCG) Before Embryo Transfer on Pregnancy Outcomes in Frozen Embryo Transfer Cycles.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Emb-025
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2016-06

CONDITIONS: Infertility
Keywords: human chorionic gonadotropin (hCG), implantation rate intrauterine hCG clinical pregnancy rate frozen embryo transfer cycles
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- experimental group (Experimental): The patients who receive 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) containing either 500 IU of hCG (Choriomon®, IBSA SA, Switzerland) is injected intrauterine, approximately 7 minutes before embryo transfer.
  Interventions: Drug: Intra uterine injection of tissue culture medium containing HCG+ET
- placebo group (Placebo Comparator): The patients who receive only 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) is injected intrauterine, approximately 7 minutes before embryo transfer.
  Interventions: Drug: Intra uterine injection of tissue culture medium +ET
- control group (Other): The patients for whom the embryonic transfer is done without the intrauterine hCG injection. The ET procedure is performed just like in the other two groups
  Interventions: Procedure: ET

INTERVENTIONS:
Drug: Intra uterine injection of tissue culture medium containing HCG+ET — 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) containing either 500 IU of hCG (Choriomon®, IBSA SA, Switzerland) is injected intrauterine, approximately 7 minutes before embryo transfer.
  Arms: experimental group
Drug: Intra uterine injection of tissue culture medium +ET — ) only 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) is injected intrauterine, approximately 7 minutes before embryo transfer.
  Arms: placebo group
Procedure: ET — the embryo transfer ( ET) is done without the intrauterine hCG injection. The ET procedure is performed just like in the other two groups.
  Arms: control group

SUMMARY:
The present study is designed as a pilot study with 50 patients in each group. Data collection form will be filled by the researcher who does not know the type of intervention in each group

DETAILED DESCRIPTION:
This randomized double blinded clinical trial is conducted to evaluate the effect of intrauterine injection of human chorionic gonadotropin (hCG) before frozen embryo transfer (ET). The study protocol is approved by the Ethics Committee (Institutional Review Board) of Royan institute. The study is performed according to the Declaration of Helsinki for medical research. All participants provide informed consent after explaining the purpose of the study. All the patients with primary infertility who have only one fresh implantation failure and undergoing frozen embryo transfer cycles are enrolled. In all patients, endometrial preparation is performed by hormonal replacement method. In this way, endometrial preparation is started from the second or third day of menstrual cycle with daily administration of 6 mg oral estradiol valerate (Estraval®, Aburaihan CO, Tehran, Iran) for 8 days. After 8 days of estradiol administration, if favourable thickness of endometrium (≥ 8 mm) is confirmed by ultrasound, estradiol valerate is continued with the same dose and 50 mg progesterone (Progestin®, Aburaihan Pharmaceutical. Co., Tehran, Iran) intramuscularly is administered for 3 days and then embryos are transferred. Otherwise the dosage of estradiol is increased to 8 mg/day until the favourable thickness of endometrium be achieved. In the Embryo transfer day, the eligible patients are randomized using sealed opaque envelopes into three groups. In all study groups, the patient is put in the lithotomy position, and the cervix is visualized using Cusco's speculum. The cervical mucous is wiped out using a sterile piece of gauze, and then the mucous is partially removed by gentle suction with a 1-mL syringe. Embryo transfer is performed using a soft catheter (Labotec, Gottingen Germany). After the catheter is passed the internal cervical os; in group A (experimental group) 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) containing either 500 IU of hCG (Choriomon®, IBSA SA, Switzerland) is injected intrauterine. In group B (the placebo group) only 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) is injected intrauterine. In both groups, approximately 7 minutes after injection, the embryos are loaded into another ET catheter and are transferred into the uterine cavity. In group C (the control group), the ET is done without the intrauterine hCG injection. The ET procedure is performed just like in the other two groups.

According to the patients' age, up to 3 frozen-thawed Embryos are thawed and transferred at cleavage stage. Hormone therapy is continued until pregnancy test (2 weeks after ET) is performed and in case of positive pregnancy, administration of estradiol valerate and progesterone continued by 10 and 12 weeks of gestation. Chemical pregnancy is defined by a rising hCG level in serum without the detection of a gestational sac. Clinical pregnancy is diagnosed by the presence of a gestational sac with fetal heart in vaginal ultrasonography. The miscarriage rate is defined as the loss of pregnancy before 20 weeks' gestational age.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of one fresh embryo transfer failure
2. Patients with Primary infertility
3. Patients with at least one embryo with excellent quality

Exclusion Criteria:

1. Female age over 40 years old
2. Severe male factor (Azoospermia)
3. Endometriosis diagnosis and the presence of hydrosalpinges
4. Uterine factor ( polyps, myoma and previous myomectomy, …)
5. Patients with polycystic ovarian syndrome diagnosis
6. Cases with pre-implantation genetic diagnosis (PGD)indication
7. Cases with difficult embryo transfer or use of Tenaculum
8. Patients with repeated implantation failures and repeated miscarriages.
9. Female smokers

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 6 weeks
  Evaluation of Implantation rate 6 weeks after embryo transfer.

SECONDARY OUTCOMES:
Pregnancy loss | 12 weeks
  Evaluation of pregnancy loss under 12 weeks of gestational age.
Early miscarriage rate | 12 weeks
  Evaluation of Early miscarriage rate under 12 weeks of gestational age.
Late miscarriage rate | 20 weeks
  Evaluation of late miscarriage rate under 20 weeks of gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahere Madani, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Maryam Hafezi, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Arezoo Arabipour, M.S.c, Principal Investigator — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://royaninstitute.org
- See also: Publication — https://doi.org/10.1007/s00404-018-4752-2